CLINICAL TRIAL: NCT02892240
Title: Retrospective Evaluation of Total Hip Replacement After Acetabular Fractures
Acronym: PTHPOSTCOTYL
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PTHPOSTCOTYL
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Total Hip; Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention. Observational study

SUMMARY:
In 1965, Emile Letournel and Robert Judet reported their experiences on acetabular fractures at the 5th day of the Raymond Poincaré Hospital in Garches. Classification Letournel is still relevant and in use today.

Many studies have sought to determine if the treatment had to be surgical or orthopedic. Although the standard treatment of displaced fractures of the acetabulum is the reduction and osteosynthesis, some advocate the THA in elderly patients with comminuted fracture of the acetabulum, impaction of the femoral head or acetabular impaction affecting more than 40% of the articular surface and including bearing zone. All these treatments and those supported have been studied in the literature.

However the study of the laying of total hip remote trauma after acetabular fracture osteosynthesis or treated conservatively, is not rich in literature. Only a few articles have been published in recent years.

Indeed, a recent review of the literature are nearly 11 series focusing on the results remotely hip prostheses for treatment of acetabular fracture. These two prospective series with between 21 and 63 patients. All authors report rates well above those reported complications for primary arthroplasty, with a revision of rates ranging between 0 and 26.5%.

Fractures of the acetabulum are covered in our service by one operator using the same release technique based on the stiffening. The objective of this study is to determine whether the systematic surgical treatment of these patients by an experienced operator reduces the high complication rate.

DETAILED DESCRIPTION:
II. objectives:

1. Evaluation of the rate and type of complications intraoperative and postoperative, and revision rates.
2. Evaluation of clinical results based on surgical strategies.

III. Methodology

This is a single-center retrospective study single-operator regarding the evaluation of surgical practice cited in goal.

Patients were aware of the potential use of their data for medical research through oral information provided by the doctor at the signing by the patient's consent related to the surgery.

IV. Nature of the data collected

The data is anonymous and unidentifiable.

Data collected include:

* The characteristics of the patient, as well as its history,
* The particular technical operating data,
* The nature of possible post-operative complications
* The clinical and radiological assessment at follow: AP pelvic radiograph, Harris score and score Postel Merle D'aubigné.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a fracture of the acetabulum ostéosynthèsée treated conservatively or who had a total hip replacement by secondary intention.
* Operated at St. Joseph's Hospital between 2005 and 2013
* Decline minimum of one year.

Exclusion Criteria:

• Total first-line hip arthroplasty following fracture of the acetabulum made within two months following the date of the initial trauma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had a fracture of the acetabulum ostéosynthèsée treated conservatively or who had a total hip replacement by secondary intention, operated at St. Joseph's Hospital between 2005 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the success of the surgical strategy | month 6
  According to the surgery strategy adopted, the investigators will response to the simple question. Success or not success?

CONTACTS AND LOCATIONS:
Overall Officials: Pomme P JOUFFROY, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided